CLINICAL TRIAL: NCT03891537
Title: Evaluation Of The Neural Therapy Effect On Long Term Postoperative Discomforts İn Patients Who Undergo Bilateral Tubal Ligation
Brief Title: Neural Therapy Effect and Bilateral Tubal Ligation
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, principal investigator, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.10.36
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Tubal Obstruction; Dysmenorrhea
Keywords: Bilateral Tubal Ligation; Postoperative Discomforts
MeSH Terms: conditions — Fallopian Tube Diseases; Dysmenorrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the effect of nebulisation in patients with bilateral tubal ligation in the first postoperative year, the amount of dysmenorrhea, dyspareunia and menstrual bleeding, recurrent vaginitis and cystitis.

A retrospective analysis of bilateral tubal ligation with optional modified Pomeroy technique in the family planning unit and evaluation of the results of patients who underwent Neural Therapy during and postoperatively will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent bilateral tubal ligation with modified Pomeroy technique,
* Patients with dysmenore, dyspareunia and menstrual bleeding,

Exclusion Criteria:

* postoperative asymptomatic
* Additional treatments for pain and complaints

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who had bilateral tubal ligation with modified Pomeroy technique and had complaints such as dysmenorrhea dyspareunia in the first postoperative year
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
postoperative dysmenorrhea | 1st year postoperative
  Postoperative dysmenorrhea in the first postoperative year was evaluated by viscous pain scale (VAS) in patients who underwent bilateral tubal ligation with the modified Pomeroy technique. There is no pain at zero points according to visuel pain scale;Ten points are very severe - unbearable pain.
  patients will score between one to ten pains.
postoperative dyspareunia | 1st year postoperative
  Postoperative dyspareunia in the first postoperative year was evaluated by viscous pain scale (VAS) in patients who underwent bilateral tubal ligation with the modified Pomeroy technique. There is no pain at zero points according to visuel pain scale;Ten points are very severe - unbearable pain.
  patients will score between one to ten pains.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)